CLINICAL TRIAL: NCT02922647
Title: Suprapubic Versus Transurethral Catheterization After Rectal Resection With Low Anastomosis for Cancer in Males
Acronym: GRECCAR10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC14.457
Record Dates: First submitted 2016-02-04; First posted 2016-10-04 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Infection; Cancer
MeSH Terms: conditions — Infections; Neoplasms | interventions — Cystostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- suprapubic catheterization (Experimental): Intervention:suprapubic catheterization after rectal resection with low anastomosis. Evaluate the urinary tract infection rate on the four days postoperative.
  Interventions: Device: suprapubic catheterization
- transurethral catheterization (Active Comparator): Intervention:transurethral catheterization after rectal resection with low anastomosis. Evaluate the urinary tract infection rate on the four days postoperative.
  Interventions: Device: transurethral catheterization

INTERVENTIONS:
Device: suprapubic catheterization — Experimental Arm: Suprapubic catheterization after rectal resection with low anastomosis for cancer in males
  Arms: suprapubic catheterization
Device: transurethral catheterization — Active comparator: Transurethral catheterization after rectal resection with low anastomosis for cancer in males
  Arms: transurethral catheterization

SUMMARY:
The purpose of this study is to compare the urinary tract infection rate on the four postoperative day between the 2 groups of patients who have undergone total mesorectal excision for cancer and low anastomosis, with either suprapubic or transurethral catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Male patients of at least 18 years of age
* Histologically proven rectal adenocarcinoma
* Stage T1-4 Nx Mx
* With or without neoadjuvant treatment
* TME and low anastomosis (colorectal or coloanal, stapled or handsewn)
* With or without loop ileostomy
* Open or laparoscopic approach
* Patient and doctor have signed a study specific informed consent form

Exclusion Criteria:

* Colonic and upper third rectal cancer (No or Partial Mesorectal Excision)
* Abdominoperineal resection
* Associated prostate, and/or seminal glands and/or bladder resection
* Infected tumour, Emergency surgery
* Epidural analgesia
* Patient with antibiotic therapy (other than prophylaxis)
* Previous treated/untreated known prostate or bladder carcinoma
* Patient with symptomatic preoperative voiding dysfunction (IPSS score >19)
* Medical history of bladder catheterization for obstruction, or urethral surgery
* Patient necessitating urinary output monitoring (impaired renal function etc)
* Patient deprived of liberty or under guardianship or incapable of giving consent
* Against the usual indications of suprapubic drainage and / or urethral sounding any known allergies to medical device materials. (p. ex. latex) and in general the known allergies to sterilizing agents (particularly oxide ethylene and its derivatives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-10-14; Primary Completion 2020-05-18 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Number of participants with urinary tract infection when using suprapubic versus transurethral catheterization as assessed by significant bacteriuria and pyuria | four days postoperative
  The urinary tract infection, defined as significant bacteriuria ( > 104 CFU / mL) and pyuria (> 6 white blood cells per high power field) in urine samples obtained immediately after removal of the urethral catheter or clamping suprapubic catheter and removing the fourth postoperative day.

SECONDARY OUTCOMES:
Duration of catherism as assessed by the number of days for participants with the catheter and number of participants leaving the hospital with the catheter | 1 month
Pain as assessed by visual analogue scale (0 to 10 score) for abdomen and urethra | at 1, 2, 3 and 4 days
  visual analogue scale (0-10) for both the abdomen and the urethra (a measure daily until hospital discharge )
Participants morbidity and mortality as assessed by Dindo and Clavien classification | at 1 month and 6 months
Rate of satisfaction for participants as assessed by questionnaries (Fact-C and EQ-5D-3L | at 30 days and 6 months
  Patient satisfaction : very, or moderately dissatisfied , unchanged , slightly , moderately , or very disappointed at the exit of the Fact- C hospital and EQ-5D - 3L at 30 days and 6 months.
Cost as assessed by the addition of the costs of the full process depending on the catheterism duration and additional consultations and readmissions for complications | at 6 months
  Estimated cost of complications, urologic surgery, medication , hospitalization, additional consultations and readmissions.
Duration of hospital stay in days | within 6 months
  the hospital stay by day
Rate of recatheterization | in the first 6 months
Duration of postoperative return to normal bladder function as assessed by IPSS score | at 1 and 6 months
Number of additionnal consultations | in the first 6 months
Lack of comfort as assessed by visual analogue scale (0 to 10 score) for abdomen and urethra | at 1, 2, 3 and 4 days
  visual analogue scale (0-10) for both the abdomen and the urethra (a measure daily until hospital discharge )
Specific complications | in the first 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pr Jean Luc FAUCHERON, Principal Investigator — University Clinic of Digestive Surgery and Emergency
Locations (1):
- University Hospital Grenoble, Grenoble, Auvergne-Rhône-Alpes, France

REFERENCES:
- [Background] Shah EF, Huddy SP. A prospective study of genito-urinary dysfunction after surgery for colorectal cancer. Colorectal Dis. 2001 Mar;3(2):122-5. doi: 10.1046/j.1463-1318.2001.00221.x. PMID 12791005
- [Background] Sterk P, Shekarriz B, Gunter S, Nolde J, Keller R, Bruch HP, Shekarriz H. Voiding and sexual dysfunction after deep rectal resection and total mesorectal excision: prospective study on 52 patients. Int J Colorectal Dis. 2005 Sep;20(5):423-7. doi: 10.1007/s00384-004-0711-4. Epub 2005 Apr 22. PMID 15846498
- [Background] Branagan GW, Moran BJ. Published evidence favors the use of suprapubic catheters in pelvic colorectal surgery. Dis Colon Rectum. 2002 Aug;45(8):1104-8. doi: 10.1007/s10350-004-6368-9. PMID 12195198
- [Background] Lee SY, Kang SB, Kim DW, Oh HK, Ihn MH. Risk factors and preventive measures for acute urinary retention after rectal cancer surgery. World J Surg. 2015 Jan;39(1):275-82. doi: 10.1007/s00268-014-2767-9. PMID 25189452
- [Background] Platt R, Polk BF, Murdock B, Rosner B. Mortality associated with nosocomial urinary-tract infection. N Engl J Med. 1982 Sep 9;307(11):637-42. doi: 10.1056/NEJM198209093071101. PMID 7110215
- [Background] Tambyah PA, Oon J. Catheter-associated urinary tract infection. Curr Opin Infect Dis. 2012 Aug;25(4):365-70. doi: 10.1097/QCO.0b013e32835565cc. PMID 22691687
- [Background] Rasmussen OV, Korner B, Moller-Sorensen P, Kronborg O. Suprapubic versus urethral bladder drainage following surgery for rectal cancer. Acta Chir Scand. 1977;143(6):371-4. No abstract available. PMID 605738
- [Background] Shapiro J, Hoffmann J, Jersky J. A comparison of suprapubic and transurethral drainage for postoperative urinary retention in general surgical patients. Acta Chir Scand. 1982;148(4):323-7. PMID 7136436
- [Background] Sethia KK, Selkon JB, Berry AR, Turner CM, Kettlewell MG, Gough MH. Prospective randomized controlled trial of urethral versus suprapubic catheterization. Br J Surg. 1987 Jul;74(7):624-5. doi: 10.1002/bjs.1800740731. PMID 3304522
- [Background] Piergiovanni M, Tschantz P. [Urinary catheterization: transurethral or suprapubic approach?]. Helv Chir Acta. 1991 Jul;58(1-2):201-5. French. PMID 1938446
- [Background] O'Kelly TJ, Mathew A, Ross S, Munro A. Optimum method for urinary drainage in major abdominal surgery: a prospective randomized trial of suprapubic versus urethral catheterization. Br J Surg. 1995 Oct;82(10):1367-8. doi: 10.1002/bjs.1800821024. PMID 7489167
- [Background] Ratnaval CD, Renwick P, Farouk R, Monson JR, Lee PW. Suprapubic versus transurethral catheterisation of males undergoing pelvic colorectal surgery. Int J Colorectal Dis. 1996;11(4):177-9. doi: 10.1007/s003840050038. PMID 8876274
- [Background] Perrin LC, Penfold C, McLeish A. A prospective randomized controlled trial comparing suprapubic with urethral catheterization in rectal surgery. Aust N Z J Surg. 1997 Aug;67(8):554-6. doi: 10.1111/j.1445-2197.1997.tb02037.x. PMID 9287924
- [Background] Baan AH, Vermeulen H, van der Meulen J, Bossuyt P, Olszyna D, Gouma DJ. The effect of suprapubic catheterization versus transurethral catheterization after abdominal surgery on urinary tract infection: a randomized controlled trial. Dig Surg. 2003;20(4):290-5. doi: 10.1159/000071693. Epub 2003 Jun 5. PMID 12789024
- [Background] McPhail MJ, Abu-Hilal M, Johnson CD. A meta-analysis comparing suprapubic and transurethral catheterization for bladder drainage after abdominal surgery. Br J Surg. 2006 Sep;93(9):1038-44. doi: 10.1002/bjs.5424. PMID 16804872
- [Background] Niel-Weise BS, van den Broek PJ. Urinary catheter policies for short-term bladder drainage in adults. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD004203. doi: 10.1002/14651858.CD004203.pub2. PMID 16034924
- [Background] Healy EF, Walsh CA, Cotter AM, Walsh SR. Suprapubic compared with transurethral bladder catheterization for gynecologic surgery: a systematic review and meta-analysis. Obstet Gynecol. 2012 Sep;120(3):678-87. doi: 10.1097/AOG.0b013e3182657f0d. PMID 22914481
- [Derived] Trilling B, Tidadini F, Lakkis Z, Jafari M, Germain A, Rullier E, Lefevre J, Tuech JJ, Kartheuser A, Leonard D, Prudhomme M, Piessen G, Regimbeau JM, Cotte E, Duprez D, Badic B, Panis Y, Rivoire M, Meunier B, Portier G, Bosson JL, Vilotitch A, Foote A, Caspar Y, Rouanet P, Faucheron JL; GRECCAR study Group. Suprapubic versus transurethral catheterization for bladder drainage in male rectal cancer surgery (GRECCAR10), a randomized clinical trial. Tech Coloproctol. 2024 Jul 2;28(1):77. doi: 10.1007/s10151-024-02950-2. PMID 38954131